CLINICAL TRIAL: NCT04331444
Title: Steno2tech CGM-The Effect of Real-time Continuous Glucose Monitoring vs. Self-monitoring of Blood Glucose on Glycemic Variables and Patient Reported Outcomes in Adults With Type 2 Diabetes Treated With Insulin-A Randomized Controlled Trial.
Brief Title: Steno2tech - Continuous Glucose Monitoring and Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Nanna Lind, RN, MSc. in nursing, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Steno2tech CGM
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; Continuous glucose monitoring; Insulin-treated; RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A, CGM (Experimental): Addition of a calibration free real-time CGM in 12 months in persons with type 2 diabetes treated with insulin.
  The participants will participate in a training course that will include the influence of different food items and exercise on glucose levels, how to measure SMBG correctly. Furthermore, participants in group A (intervention) will, in similarity to the HCPs, receive a CGM-education and training session led by the study investigator and will be interactive and hands-on, using case studies. The training session will include spoken and written instructions on how to insert and wear the CGM device and how to interpret the CGM information to better understand the relation between participants blood glucose and their diabetes self-management.
  Interventions: Device: CGM; Behavioral: training course
- Group B, CGM + peer-support (Experimental): Addition of a calibration free real-time CGM in 12 months in persons with type 2 diabetes treated with insulin plus 3 sessions of peer-support in groups of 6 participants.
  The participants will participate in a training course that will include the influence of different food items and exercise on glucose levels, how to measure SMBG correctly. Furthermore, participants in group B (intervention incl. peer-support) will, in similarity to group A, receive a CGM-education and training session. The training and CGM-course for participants in group B are similar to the course for group A with the addition of three peer-support sessions. The approach will be participatory and adaptable to allow flexibility in the content of the peer-support sessions and involving customized use of participatory methods i.e. dialogue tools and exercises.
  Interventions: Device: CGM; Behavioral: training course; Behavioral: Peer-support
- Group C, SMBG (Active Comparator): Standard self-monitoring of blood glucose according to standard guidelines, in 12 months.
  The participants will participate in a training course that will include the influence of different food items and exercise on glucose levels, how to measure SMBG correctly.
  Interventions: Behavioral: training course

INTERVENTIONS:
Device: CGM — Using the CGM during the entire study period of 12 months.
  Other Names: Continuous glucose monitoring
  Arms: Group A, CGM; Group B, CGM + peer-support
Behavioral: training course — The participants in the three groups will attend a three-hour training course with different content depending on the group allocation. The aim of this training course is to ensure that the participants have the knowledge, support and confidence to work collaboratively with their HCPs to increase TIR and decrease HbA1c.
Behavioral: Peer-support — The peer-support will be facilitator-led by the primary investigator with peer exchange in group sessions (3 sessions over the study period, 3 hours per session) with 6-8 participants in every group.
  Other Names: Group sessions
  Arms: Group B, CGM + peer-support

SUMMARY:
The overall objective of this research study is to examine the effectiveness of the use of CGM vs. SMBG in persons with insulin-treated type 2 diabetes on glycemic variables and patient reported outcomes on treatment satisfaction, health behavior and wellbeing. The independent effect of peer-support will also be studied.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes is increasing. Although medical treatment options have increased, still less than a third obtain their optimal glycemic goal. The use of continuous glucose monitoring (CGM) in persons with type 1 diabetes has shown to be the most important driver for improvement in glycemic control-even more than insulin-pump therapy-but the use of technology in type 2 diabetes are not yet reimbursed and has been investigated in very few studies.

The study will be a single center, prospective, randomized, open-labelled, three-armed study with the randomization 2:1:2 in group A with CGM, group B with CGM and peer-support, group C as a control group with SMBG. The study will run for 12 months and will include 100 adult participants with insulin-treated type 2 diabetes, treated at the outpatient clinic at Steno Diabetes Center Copenhagen. Recruitment will begin in August 2020 and end in May 2022. Final 12-month follow-up is anticipated to be in July 2023.

The study is investor-initiated. The primary investigator (Nanna Lind, PhD. Student) will be responsible for execution of this study under guidance by the sponsor Kirsten Nørgaard. Results will be published in international peer-reviewed journals.

Our study will provide evidence of the effectiveness of the use of CGM in the treatment for type 2 diabetes, potentially shaping clinical guidelines for SMBG frequency and timing as well as use of technology in type 2 diabetes with an impact on both healthcare and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes according to clinical definitions
* Treated with insulin injections at least once daily on top of diet and exercise recommendations. Insulin therapy has been used for at least 12 months. Can be additionally treated with one or more different oral antidiabetic drugs (except sulfonylurea), and/or glucagon-like-peptide 1 (GLP-1) analogues
* Attending the outpatient clinic at Steno Diabetes Center Copenhagen for at least 12 months
* Age ≥ 18 years
* HbA1c > 58 mmol/mol (7.5%) at two consecutively measurements over at least 3 months
* Willing to use possible interventions; to perform self-monitoring of blood glucose (SMBG) as requested by the investigators AND to use CGM continuously without calibration for a 12-month period.
* Willing to intensify non-medical and medical treatment to achieve better glucose control.

Exclusion Criteria:

* Inability to understand the patient information and give informed consent
* Not speaking and understanding Danish
* Treatment with sulfonylurea (SU) during the last 3 months before study start
* New antidiabetic treatment the last three months
* Use of systematic corticosteroids
* Visual impairment
* Severe skin allergy for adhesive tape to the patch of CGM or other skin condition that inhibits the use of a CGM device
* Comorbidity which does not allow lowering of HbA1c to 53 mmol/mol (7.0%)
* Hypoglycemic unawareness
* Impaired renal disease with eGFR < 45 ml/min/1.73m2
* Conditions that impact the stability of a HbA1c measurement (chronic liver disease, haemoglobinopathy, anemia etc.)
* Known or suspected alcohol or drug abuse
* Already using Flash glucose monitoring (Libre) or CGM
* Enrolled in another clinical study
* Pregnancy, intend to become pregnant, breastfeeding or not using adequate contraceptive methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Difference between change in TIR (3.9-10 mmol/l) in percent, assessed via blinded CGM device, between CGM group (A) and SMBG group (C) | from baseline to 12 months
  Percent

SECONDARY OUTCOMES:
Difference between change in HbA1c between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  mmol/mol
Difference between change in mean sensor glucose concentration measured by 2 weeks blinded CGM between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  mmol/l
Difference between change in time below range (TBR) (< 3.9 mmol/l, < 3.0 mmol/l), in percent, measured by 2 weeks blinded CGM between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  Percent
Difference between change in time above range (TAR) (>10 mmol/l, > 13.9 mmol/l), in percent, measured by 2 weeks blinded CGM, between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  Percent
Difference between change in glycemic variability (SD, Coefficient of variance and others), measured by 2 weeks blinded CGM between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  Percent
Difference between change in number of severe hypoglycemic episodes between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  number
Difference between change in insulin dose between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  units
Difference between change in BMI between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  weight and height will be combined to report BMI in kg/m^2
Difference between change in antidiabetic medicine between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  (new medication, change in doses, discontinuation of medicine)
Difference between change in patients related outcome measures on general wellbeing, between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the questionnaire WHO-5
Difference between change in patients related outcome measures on diabetes-related distress, between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Diabetes Distress Scale
Difference between change in patients related outcome measures on hypoglycemia fear between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the short form Hypoglycemia Fear Survey
Difference between change in patients related outcome measures on diabetes treatment satisfaction between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Diabetes Treatment Satisfaction Quenstionnaire
Difference between change in patients related outcome measures on satisfaction with glucose monitor between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Glucose Monitoring Satisfaction Scale
Difference between change in health behavior regarding exercise between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Swedish National Board of Health and Welfare questionnaire for Physical Activity
Difference between change in health behavior regarding diet between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Danish Perceived Dietary Adherence questionnaire
Difference between change in health behavior regarding anti-diabetic medication adherence between the CGM group (A) and the SMBG group (C) | from baseline to 12 months
  measured by the Danish Medical Adherence Scale
Difference between change in TIR, assessed by 2 weeks blinded CGM device, and HbA1c between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  Percent
Difference between change in general wellbeing between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the questionnaire WHO-5
Difference between change in diabetes-related distress between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Diabetes Distress Scale
Difference between change in hypoglycemia fear between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the short form Hypoglycemia Fear Survey
Difference between change in glucose monitoring satisfaction between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Glucose Monitoring Satisfaction Scale
Difference between change in diabetes treatment satisfaction between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Diabetes Treatment Satisfaction Quenstionnaire
Difference between change in health behavior regarding exercise between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Swedish National Board of Health and Welfare questionnaire for Physical Activity
Difference between change in health behavior regarding diet between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Danish Perceived Dietary Adherence questionnaire
Difference between change in health behavior regarding anti-diabetic medication adherence between the CGM groups (without peer-support group A and with peer-support group B) | from baseline to 12 months
  measured by the Danish Medical Adherence Scale
Difference in mean number of days of CGM use between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  days
Difference in HbA1c baseline between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  mmol/mol
Difference in age between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  in years
Difference in diabetes duration between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  in years
Difference in C-peptide between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  pmol/l
Difference in education level between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  Percent
Difference in social status between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  measured by civil status and occupation
Difference in ethnicity between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  white/non-white
Difference in medicine used between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
Difference in change in health behavior regarding to diet between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  measured by the Danish Perceived Dietary Adherence questionnaire
Difference in change in health behavior regarding to exercise between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  measured by the Swedish National Board of Health and Welfare questionnaire for Physical Activity
Difference in change in health behavior regarding to medication adherence between individuals achieving TIR> 70% vs TIR< 70% within the CGM groups (group A+B) | from baseline to 12 months
  measured by the Danish Medical Adherence Scale
Correlation between mean number of SMBG/day and time points for SMBG in the study period and improvement in HbA1c, in TIR, in TBR, in TAR within the control group C | from baseline to 12 months
Difference between number of participants using CGM vs. not using CGM increasing 5 % or more in TIR | from baseline to 12 months
  number

OTHER OUTCOMES:
Evaluating which blood glucose measured by SMBG best reflect TIR | from baseline to 12 months
  (fasting, pre-prandial or postprandial)

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Lind, RN MSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
Study results, positive, negative and inconclusive findings, will be presented at national and international scientific meetings and published in at least three scientific papers in international scientific peer-reviewed journals and through the PhD thesis. After conclusion of the study, a final report will be generated and sent to the Regional Scientific Ethics Committee (RVK). The study protocol will furthermore be published at www.clinicaltrial.gov.

REFERENCES:
- [Derived] Lind N, Lindqvist Hansen D, Saetre Rasmussen S, Norgaard K. Real-time continuous glucose monitoring versus self-monitoring of blood glucose in adults with insulin-treated type 2 diabetes: a protocol for a randomised controlled single-centre trial. BMJ Open. 2021 Jan 15;11(1):e040648. doi: 10.1136/bmjopen-2020-040648. PMID 33452188